CLINICAL TRIAL: NCT00011557
Title: Functional Magnetic Micturition in Patients w/SCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1747R
Record Dates: First submitted 2001-02-22; First posted 2001-02-26 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2001-01

CONDITIONS: Spinal Cord Injury
Keywords: Bladder, electromagnetic fields, Spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Insemination, Artificial, Heterologous

INTERVENTIONS:
Device: Assistance in Voiding

SUMMARY:
This project will determine the ultimate usefulness of functional magnetic stimulation (FMS) as an assistive device for voiding in patients with SCI.

DETAILED DESCRIPTION:
Investigators intend to determine the ultimate usefulness of functional magnetic stimulation (FMS) as an assistive device for voiding in patients with SCI.

Thirty six persons will be recruited and will undergo an 8 week protocol for conditioning of the bladder. The investigators propose to: investigate the changes in bladder function in response to long-term bladder conditioning by FMS; further optimize the FMS technology and parameters for effective bladder emptying in SCI; evaluate the role of the external sphincter muscle fatigue by FS in facilitating bladder emptying; critically evaluate the relative response of FMS data to existing information using functional electrical stimulation;further develop criteria that will be used to predict which SCI patients are optimally suitable for FMS; establish a comprehensive stimulation criteria that will reflect the safety and effectiveness of structures associated with the bladder that are exposed to the electro-myographic field.

ELIGIBILITY:
Patients with SCI above T10 level, six months post injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 1998-01; Study Completion 2000-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fryer, Ph.D. Asst. Director — Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service; Nancy Rocheleau, Program Analyst — Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service
Locations (1):
- VAMC, Long Beach, Long Beach, California, United States